CLINICAL TRIAL: NCT04708431
Title: Androgen Receptor, Implications for Health and Wellbeing: Natural History Study of Individuals With Androgen Insensitivity
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200165; 20-CH-0165
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12-23

CONDITIONS: Androgen Insensitivity Syndrome; Metabolic Parameters in AIS, CAIS, PAIS and MAIS; Tumor Formation in AIS, CAIS, PAIS and MAIS; Sexual Function AIS, CAIS, PAIS and MAIS
Keywords: Androgen insensitivity syndrome (AIS); Complete androgen insensitivity (CAIS); Partial androgen insensitivity (PAIS); Mild androgen insensitivity syndrome (MAIS); Natural History
MeSH Terms: conditions — Androgen-Insensitivity Syndrome; Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Female subjects relatives who are carriers of the AR gene difference: We will enroll 50 female subjects relatives AIS subjects who are carriers of the AR gene difference
- Female subjects relatives who are not carriers of the AR gene: We will enroll 50 female subjects relatives of AIS subjects who are not carriers of the AR gene.
- Healthy male subjects relatives: We will enroll 50 healthy male subjects of AIS relative subjects
- Subjects with androgen receptor mutations: 500 Subjects with confirmed androgen receptor mutations

SUMMARY:
Background:

Androgen effects in humans are usually (but not always) mediated by the androgen receptor which is coded for by the androgen receptor gene (AR gene). Androgen Insensitivity Syndrome (AIS) is a rare condition in which the body cannot sense the male hormones in the blood or tissue. Both women and men can be affected by AIS. Researchers want to learn more about the health of people with AIS over time.

With a natural history study in individuals with AIS, data and tests may provide information regarding health risks (including the risks and benefits of gonadectomy and best ways to monitor for tumor) and optimal management of individuals with AIS as well as elucidate the role of the androgen receptor in human health. This study does not involve any interventions and we can provide clinical care while collecting data.

Objective:

The objective of this natural history study is to describe and define a comprehensive phenotype (characteristic) of patients with AIS based on confirmed androgen receptor (AR) gene difference. We will evaluate hormones, bone density and markers, cardiovascular and metabolic parameters, as well as quality of life and tumor formation risk and evaluation. The purpose is to obtain a better understanding of the overall health issues that people with AIS may have through the study procedures listed.

Eligibility:

People ages 0-99 with AIS and their adult relatives

Design:

Participants will go through a series of study procedures for data and specimen collection. This will be done to understand how AIS affects individuals since the androgen receptor is found in many tissues in the body including skin, bone, muscle, and the neurologic, immune and metabolic systems. All tests will be performed by skilled and trained study professionals.

Participants will be screened with:

Medical history

Physical exam

Medical record review

Lab tests.

Participants will have physical exams. Their body measurements will be taken. They will have blood and urine tests. They will have electrocardiograms to check heart health. They may complete questionnaires. They may have an Oral Glucose Tolerance Test.

Participants may have x-rays and HRpQCT scans taken of the hand, wrist, and other bones.

Participants will have body scans to measure bone thickness.

Participants will have magnetic resonance imaging (MRI) or sonogram of the pelvis. For MRI, they may get a contrast agent via intravenous (IV) catheter.

Adult participants may have the following:

MR elastography. It uses MRI and low-frequency vibrations to map stiffness of body tissues.

MR spectroscopy. It uses MRI to take pictures of chemicals in the liver and body fat.

Cardiac computed tomography scan. It uses x-rays to make pictures of the heart. Participants may get a contrast agent via IV.

Optional genital exam.

Participants will have visits every 1-2 years. Participation lasts indefinitely.

Adult relatives will also be invited to participate but will have only 1 visit. It will include some of the above tests.

DETAILED DESCRIPTION:
Study Description: This is a natural history study of individuals with androgen receptor gene abnormalities.

Objectives:

Primary Objectives:

To define and describe a comprehensive phenotype of patients with androgen insensitivity (based on confirmed androgen receptor

(AR) gene difference), including hormonal, metabolic, immunologic, and cardiovascular aspects of AIS, as well as quality life and tumor formation risk and evaluation.

Secondary Objectives:

1. Bone Health:

   - Follow a large population of patients with androgen receptor abnormalities for:
   * Longitudinal assessment of bone mineral density (BMD) before and after gonadectomy
   * Development of normative values for dual-energy X-ray absorptiometry (DEXA) and high-resolution peripheral quantitative computed tomography (HRpQCT) scans in individual with complete androgen insensitivity syndrome (CAIS) and family members.
   * Studies to determine bone geometry, strength and shape,

     * Studies to determine muscle-skeletal unit inferences
     * Studies to evaluate skin tone
   * Evaluation of bone accrual from infancy to adolescence
2. Metabolic and Immune Abnormalities:

   - Follow a large population of patients with androgen receptor abnormalities for studies of metabolic abnormalities and auto-immune disease screening
   * Metabolic syndrome,

     * Insulin resistance
     * Cardiovascular markers
     * Endometabolic imaging
   * Autoimmune screening tests
3. Testicular Tumor Risk and Monitoring:

   - Follow a large population of patients with androgen receptor abnormalities in order to:

   -- Describe the typical and atypical appearance of testes on ultrasound and magnetic resonance imaging (MRI) in young individual with

   CAIS.
   * Evaluate gonadal tumor markers as a tool to assess for gonadal tumor.

     - When individuals with androgen receptor abnormalities decide to undergo gonadectomy, perform tissue evaluation in order to:
   * Investigate the pathophysiology of gonadal tumor formation
   * Assess fertility potential in testis of individual with androgen receptor abnormalities
4. Quality of Life:

   * Follow a large population of patients with androgen receptor abnormalities to characterize quality of life measures throughout the lifespan
   * Evaluate the effects of androgen receptor abnormalities on individual s sexual function. Compare sexual function in adult individuals with androgen receptor abnormalities to individual with classic congenital adrenal hyperplasia (CAH) and unaffected individual of

   similar ages.
5. Hormone Replacement:

   - Evaluate different types and delivery of hormone replacement therapy on quality of life, sexual function, bone health and metabolic parameters in individual who have undergone gonadectomy
6. Follow a sample population of relatives of individuals with androgen insensitivity syndrome (AIS) in order to assess the effects of AR gene difference carrier status phenotype including hormonal, metabolic, immunologic, quality of life, and tumor formation. Family members without AR gene abnormalities will serve as controls.

Follow a large population of patients with AIS for referral to future treatment studies.

Endpoints:

Primary Endpoint: Longitudinal evaluation of 500 individuals with AIS.

Secondary:

* DEXA and HRpQCT scans and bone metabolism markers will be evaluated longitudinally in all individuals with AIS. Additionally, these will be correlated with muscle grip and skin tone studies.
* Compare metabolic parameters in all individuals with AIS.
* Compare gonadal tissue with MRI or ultrasound in all individuals with AIS.
* Evaluate Quality of life with Quality of Life (QoL) questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for AIS subjects

In order to be eligible to participate in this study, an individual must meet all the following criteria:

1. Individuals ages 0-99 years old with known androgen insensitivity based on pathologic androgen receptor gene mutation or based on clinical diagnosis of complete androgen insensitivity (CAIS) based on 46 XY karyotype, presence of testis, absence of uterus, high testosterone without signs of virilization at birth or during puberty and/or multiple members in the family also presenting with clinical CAIS.
2. Identify as male or female
3. Patients with both complete, partial and mild androgen insensitivity are eligible
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. Ability of subject or guardian to understand and the willingness to sign and date a written informed consent document.

Inclusion Criteria for Relative of AIS subjects

1) Adult Relatives of patients with AIS

EXCLUSION CRITERIA:

Exclusion Criteria for AIS subjects

1. An individual who meets any of the following criteria will be excluded from participation in this study: Patients with other diagnosis such as partial or complete gonadal dysgenesis, 5-alpha reductase deficiency, and 46 XY. If, following a diagnostic work-up, a patient is determined to have causes for 46 XY DSD other than androgen insensitivity; they will no longer be followed on this protocol. They will have the opportunity to continue care with the team under the Data Collection Protocol or may be referred to an expert or multidisciplinary DSD team in the community.
2. Patients with significant non-endocrine medical conditions.

Exclusion Criteria for Relative of AIS subjects

1) Patients with significant non-endocrine medical conditions.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll and evaluate 500 patients with confirmed androgen receptor mutations. We will enroll 50 female relatives who are carriers of the AR gene difference and 50 female relatives who are not carriers of the AR gene and 50 healthy male relatives.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2040-02-01 (Estimated); Study Completion 2040-02-01 (Estimated)

PRIMARY OUTCOMES:
To define and describe a comprehensive phenotype in 500 patients with androgen insensitivity | End of study
  Primary Objectives: To define and describe a comprehensive phenotype of patients with androgen insensitivity (based on confirmed androgen receptor (AR) gene difference), including hormonal, metabolic, immunologic, and cardiovascular aspects of the disease, as well as quality life and tumor formation risk and evaluation

SECONDARY OUTCOMES:
Effects of hormone therapy in individuals with Androgen Insensitivity | End of study
  Evaluate different types and delivery of hormone replacement therapy on quality of life, sexual function, bone health and metabolic parameters in individuals who have undergone gonadectomy
Quality of life measures (QoL) in individuals with Androgen Insensitivity | End of study
  Quality of life questionnaires will be administered during each patient visit
Gonadal Tumor evaluation in individuals with Androgen Insensitivity | End of study
  A) MRI and Ultrasound imaging will be performed to describe the typical appearance of testes on ultrasound and magnetic resonance imaging (MRI) in young individuals with CAIS. B) Evaluate gonadal tumor markers as a tool to assess for gonadal tumor C) Gonadectomy tissue evaluation in order to: Investigate the histology and pathophysiology of gonadal tumor formation and assess the state of spermatogenesis in testis of individuals with androgen receptor abnormalities
Metabolic assessment in individuals with Androgen Insensitivity | End of study
  Metabolic parameters including laboratory evaluation as well as novel endometabolic imaging will be performed. Imaging will include MR spectography of liver fat and body composition, MR elastography for fibrosis assessment, and coronary wall imaging using CT angiography, and MRI evaluation of endothelial function to evaluate for artherosclerosis
Evaluate Bone Health in individuals with Androgen Insensitivity | End of study
  DEXA and HRpQCT scans and bone metabolism markers will be evaluated longitudinally in all individuals with AIS and family members. Comparison between family members who are carriers and non-carriers of the AR gene difference, those with mild, partial and complete androgen insensitivity will allow for evaluation of the effect of androgen receptor abnormalities on bone mineral density and growth as well as develop normative data for DEXA and HRpQCT scan interpretation in this population. Physiatry measurements will allow evaluation of muscle skeletal unit inferences.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Gomez-Lobo, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Deans R, Creighton SM, Liao LM, Conway GS. Timing of gonadectomy in adult women with complete androgen insensitivity syndrome (CAIS): patient preferences and clinical evidence. Clin Endocrinol (Oxf). 2012 Jun;76(6):894-8. doi: 10.1111/j.1365-2265.2012.04330.x. PMID 22211628
- [Background] Ahmed SF, Cheng A, Dovey L, Hawkins JR, Martin H, Rowland J, Shimura N, Tait AD, Hughes IA. Phenotypic features, androgen receptor binding, and mutational analysis in 278 clinical cases reported as androgen insensitivity syndrome. J Clin Endocrinol Metab. 2000 Feb;85(2):658-65. doi: 10.1210/jcem.85.2.6337. PMID 10690872
- [Background] Bertelloni S, Meriggiola MC, Dati E, Balsamo A, Baroncelli GI. Bone Mineral Density in Women Living with Complete Androgen Insensitivity Syndrome and Intact Testes or Removed Gonads. Sex Dev. 2017;11(4):182-189. doi: 10.1159/000477599. Epub 2017 Jul 18. PMID 28715798
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-CH-0165.html